CLINICAL TRIAL: NCT02067637
Title: Delayed Effects of Treatment in Cancer Survivors (DETECS)
Acronym: DETECS
Status: Withdrawn | Type: Observational
Why Stopped: Low accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 13-1761.cc
Record Dates: First submitted 2014-02-12; First posted 2014-02-20 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Leukemia; Lymphoma; Gynecologic Cancer
Keywords: cancer therapy, cancer treatment
MeSH Terms: conditions — Breast Neoplasms; Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed: Individuals with one of the following cancer diagnoses: breast, leukemia, lymphoma, and/or any gynecologic cancer.
- Unexposed: Healthy controls

SUMMARY:
Hypotheses and Specific Aims: There is limited data on the long-term consequences of cancer therapy on young, reproductively aged cancer survivors. The investigators objective is to characterize some of these effects in the cancer population.

DETAILED DESCRIPTION:
Specific Aim 1: To compare markers of ovarian reserve between cancer survivors and healthy controls.

Hypothesis: Cancer survivors will have lower serum Anti-Mullerian Hormone (AMH) and antral follicle count (AFC), and higher Follicle Stimulating Hormone (FSH) than healthy controls.

Specific Aim 2: To compare cardio-metabolic, endocrine and bone profiles between cancer survivors and controls using a combination of anthropometric measures, fasting serum markers, and urinary markers of bone health.

Hypothesis: Cancer survivors will have higher total cholesterol and lower 25-OH vitamin D than healthy controls.

Specific Aim 3: To evaluate potential associations between ovarian reserve and markers of metabolism, obesity, and tumor bone health in young female cancer survivors.

Hypothesis: As BMI and total cholesterol increases, serum AMH will decrease.

Specific Aim 4: To compare quality of life markers, as assessed by validated instruments, between cancer survivors and controls using recommended scoring techniques.

Hypothesis: Cancer survivors will have lower quality of life markers as compared to controls.

The investigators will conduct a prospective study to characterize the quality of life and cardio-metabolic, endocrine, and bone profiles of female cancer survivors using a combination of anthropometric, serum, urinary, and ultrasonographic markers in combination with QOL instruments.

ELIGIBILITY:
Inclusion Criteria:

* Exposed: Females between the ages of 18 and 45, at least 2 years from the completion of cancer therapy. Subjects will have one of the following cancer diagnoses: breast, leukemia, lymphoma, and/or any gynecologic cancer. Subjects must also be postmenarchal, have a uterus, at least one intact ovary, and must be willing and able to comply with study procedures. Subjects can be of any menopausal status and within 10 years post treatment.
* Unexposed: Females between the ages of 18 and 45 with no prior history of cancer treatment.

Exclusion Criteria:

* Exposed: Pregnancy, lactation within the previous 3 months, any medical condition other than cancer with a known correlation with premature menopause (i.e. Turner's syndrome, Fragile X, gonadal dysgenesis, polyglandular autoimmune syndrome, lupus, etc.), hormonal contraceptive use within 3 months.
* Unexposed: Healthy controls with a history of polycystic ovary syndrome (PCOS), diabetes, thyroid dysfunction, hypertension, and hypercholesterolemia will be excluded in addition to cancer patients or survivors with one of the aforementioned diseases diagnosed prior to cancer diagnosis or treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Prospective cohort study of female cancer survivors who are at least 2 years from completion of cancer therapy and healthy controls age less than 45 years.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Serum anti-Mullerian hormone (AMH) | Day 0 - 1 time measurement
  Test of ovarian reserve via a blood sample.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Day 0 - 1 time measurement
  Height and weight will be measured to calculate BMI.
Antral Follicle Count | Day 0 - 1 time measurement
  Measure of ovarian reserve via a transvaginal ultrasound.
Hemoglobin A1c | Day 0 - 1 time measurement
  Will measure the percentage of hemoglobin that is coated with sugar (glycated).
High sensitivity C reactive protein (hsCRP) | Day 0 - 1 time measurement
  We will measure low levels of C-reactive protein (CRP) by blood test. The test will be done to determine risk for heart disease.
Follicle-stimulating hormone (FSH) | Day 0 - 1 time measurement
  We will measure the amount of follicle-stimulating hormone (FSH) in a blood sample.
25-OH vitamin D | Day 0 - 1 time measurement
  We will measure how much vitamin D is present via a blood test.
Estrone | Day 0 - 1 time measurement
  We will measure the amount of estrone (form of estrogen) by testing a urine sample.
Pregnanediol | Day 0 - 1 time measurement
  We will measure the amount of pregnanediol by testing a urine sample. This is an indirect way to measure progesterone levels in the body.
Testosterone | Day 0 - 1 time measurement
  We will measure the amount of the steroid hormone testosterone by testing a blood sample.
Ovarian volume | Day 0 - 1 time measurement
  Ovarian volume will be measured via a transvaginal ultrasound.
Quality of Life | Day 0 - 1 time measurement
  Validated instruments will be used to compare quality of life markers between cancer survivors and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Laxmi Kondapalli, MD, MSCE, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Clinical and Translational Research Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iughetti L, Bruzzi P, Predieri B, Paolucci P. Obesity in patients with acute lymphoblastic leukemia in childhood. Ital J Pediatr. 2012 Jan 27;38:4. doi: 10.1186/1824-7288-38-4. PMID 22284631
- [Background] Landy DC, Miller TL, Lopez-Mitnik G, Lipsitz SR, Hinkle AS, Constine LS, French CA, Rovitelli AM, Adams MJ, Lipshultz SE. Aggregating traditional cardiovascular disease risk factors to assess the cardiometabolic health of childhood cancer survivors: an analysis from the Cardiac Risk Factors in Childhood Cancer Survivors Study. Am Heart J. 2012 Feb;163(2):295-301.e2. doi: 10.1016/j.ahj.2011.11.008. PMID 22305850
- [Background] Nandagopal R, Laverdiere C, Mulrooney D, Hudson MM, Meacham L. Endocrine late effects of childhood cancer therapy: a report from the Children's Oncology Group. Horm Res. 2008;69(2):65-74. doi: 10.1159/000111809. Epub 2007 Dec 5. PMID 18059086
- [Background] Sklar C, Boulad F, Small T, Kernan N. Endocrine complications of pediatric stem cell transplantation. Front Biosci. 2001 Aug 1;6:G17-22. doi: 10.2741/a714. PMID 11487479
- [Background] Gleeson HK, Shalet SM. Endocrine complications of neoplastic diseases in children and adolescents. Curr Opin Pediatr. 2001 Aug;13(4):346-51. doi: 10.1097/00008480-200108000-00011. PMID 11717561
- [Background] Toner JP, Philput CB, Jones GS, Muasher SJ. Basal follicle-stimulating hormone level is a better predictor of in vitro fertilization performance than age. Fertil Steril. 1991 Apr;55(4):784-91. doi: 10.1016/s0015-0282(16)54249-6. PMID 1901282
- [Background] Lee MM, Donahoe PK, Hasegawa T, Silverman B, Crist GB, Best S, Hasegawa Y, Noto RA, Schoenfeld D, MacLaughlin DT. Mullerian inhibiting substance in humans: normal levels from infancy to adulthood. J Clin Endocrinol Metab. 1996 Feb;81(2):571-6. doi: 10.1210/jcem.81.2.8636269.
- [Background] Di Paola R, Costantini C, Tecchio C, Salvagno GL, Montemezzi R, Perandini A, Pizzolo G, Zaffagnini S, Franchi M. Anti-Mullerian hormone and antral follicle count reveal a late impairment of ovarian reserve in patients undergoing low-gonadotoxic regimens for hematological malignancies. Oncologist. 2013;18(12):1307-14. doi: 10.1634/theoncologist.2013-0138. Epub 2013 Oct 22. PMID 24149138
- [Background] Lutchman Singh K, Muttukrishna S, Stein RC, McGarrigle HH, Patel A, Parikh B, Groome NP, Davies MC, Chatterjee R. Predictors of ovarian reserve in young women with breast cancer. Br J Cancer. 2007 Jun 18;96(12):1808-16. doi: 10.1038/sj.bjc.6603814. Epub 2007 May 29. PMID 17533402